CLINICAL TRIAL: NCT04858386
Title: The Use of Early Pregnancy HbA1c in Predicting Excessive Fetal Growth in Women at Risk of Glucose Intolerance
Acronym: SHAPE
Status: Terminated | Type: Observational
Why Stopped: Covid-19
Sponsor: Belfast Health and Social Care Trust (Other)
Collaborators: Queen's University, Belfast (Other)
Responsible Party: Sponsor
Other Study IDs: 17024UG-SW
Record Dates: First submitted 2021-04-21; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Gestational Diabetes
Keywords: HbA1c; Fetal Growth; Macrosomia; Visceral Fat; Pregnancy; Glucose Intolerance
MeSH Terms: conditions — Diabetes, Gestational; Glucose Intolerance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Frozen Serum Frozen Plasma Frozen centrifuged urine
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The association of hyperglycaemia in pregnancy (gestational diabetes mellitus; GDM) with adverse maternal and fetal outcomes is clearly recognised. Traditionally the diagnosis is made at 28 weeks gestation at which stage children of affected women already have a two-fold rate of excessive weight gain (abdominal circumference > 90th percentile). This is attributed to fetal exposure to undiagnosed high blood glucose earlier in pregnancy. Indeed almost 25% of women with GDM develop the condition before 20 weeks gestation. Interventional studies in women diagnosed in the late second trimester have shown benefits in reducing fetal macrosomia. It is unknown whether screening in the first trimester would predict fetal macrosomia and allow more timely and effective intervention. To examine this question, we propose a prospective cohort study of 1,662 women at increased risk of GDM to determine if an elevated HbA1c (39-48mmool/l) in early pregnancy (<14 weeks) can identify babies at risk of excessive weight gain in later pregnancy, as determined by ultrasound measurement of abdominal circumference at 28 weeks gestation. The study will be largely integrated into routine clinical practice enabling a large number of women to participate. Study participants will all undergo formal screening (75g oral glucose tolerance test) for GDM at 28 weeks gestation. Secondary outcomes, namely the ability of early pregnancy HbA1c to predict later maternal GDM, and fetal and maternal complications of pregnancy will also be evaluated. The results of this study, if positive, are likely to impact upon patient care almost immediately following study completion. In addition, given the stability of the Northern Ireland population, the relatively unique data set will facilitate future work on predictive markers for cardiovascular disease, and prospective studies on the cardiovascular consequences of GDM on both mother and baby.

DETAILED DESCRIPTION:
Study Aim: The overall aim of this study is to identify a feasible, easily adopted, early screening method for excessive fetal weight gain; a known risk factor for childhood obesity and type 2 diabetes.

Primary objective: To examine the effect of increased (39-48mmol/mol) maternal HbA1c, measured before 14 weeks gestation, on the ultrasound finding of fetal abdominal circumference greater than the 90th percentile at 28 weeks gestation. We hypothesise that women with a high early pregnancy HbA1c (39-48mmol/mol) will have a significantly increased risk of excessive weight gain in their babies.

Secondary objectives:

1. To establish ability of maternal HbA1c in early pregnancy (< 14 weeks) to predict the diagnosis of GDM in the late second trimester (28 weeks)
2. To determine the effect of an increased (39-48mmol/mol) maternal HbA1c, measured before 14 weeks gestation, on fetal, maternal and neonatal complications of pregnancy (stillbirth, preterm delivery, birth weight >90th percentile, shoulder dystocia, birth injury, neonatal hypoglycaemia, neonatal intensive care, caesarean delivery, preeclampsia, gestational hypertension) taking account of any GDM intervention.
3. To determine dietary patterns among women with and without a diagnosis of GDM.

Study Outline: Prospective cohort study of women at increased risk of GDM presenting for obstetric care at the Royal Jubilee Maternity Hospital Belfast; the largest maternity unit in Northern Ireland with some 5000-6000 deliveries per year. The study will be conducted over three years by healthcare staff with support from the research team. The study will largely be integrated into routine clinical practice thus enabling a large number of women to take part in the study.

Participants: 1,828 women in early pregnancy (≤ 14 weeks gestation) will be recruited, following informed consent, during their booking visit at the Royal Jubilee Maternity Hospital, Belfast. Inclusion criteria include age ≥ 18yrs, and NICE risk factors for glucose intolerance namely body mass index ≥ 30kg/m2, family history of diabetes (first-degree relative), previous macrosomic baby (>4.5kg) and minority ethnic family origin with a high prevalence of diabetes14. Exclusion criteria will include pre-existing type 1 or type 2 diabetes mellitus, a previous history of GDM, booking HbA1c ≥ 48mmol/mol (6.5%), anaemia diagnosed on booking full blood count, booking diagnosis of a multiple pregnancy, and use of corticosteroids or metformin within two weeks of booking.

Booking visit: Participants at 10-14 weeks gestation will be consented at their booking visit. At this visit patient demographics such as height, weight and blood pressure, are recorded on the Northern Ireland Maternity Information System (NIMATS) by the booking midwife. Study blood samples (14 mls) will be taken alongside routine antenatal bloods by the booking midwife, and plasma analysed for HbA1c (4mls) in the Regional Haematology Laboratory as outlined below. Serum and urine will also be collected (10mls whole blood, 10mls urine), processed and stored at -80°C for future work. Sample processing (as outlined below) will be carried out immediately following venesection/urine collection. Women with HbA1c ≥ 48mmol/mol (6.5%) will informed of their result by telephone (RD); referred for ongoing care at the Diabetes Antenatal Clinic and excluded from the study. Women with HbA1c < 48mmol/mol (6.5%) will be recruited to the study but will continue to be managed according to their routine obstetric care pathway. Women booking at the Royal Jubilee Maternity Hospital will also be offered ultrasound measurement of visceral/subcutaneous fat depth. This will be performed at the end of their routine booking ultrasound (RD) and measurements will be recorded in the study database.

Nested Observational Study In a subset of women, visceral adipose tissue depth and subcutaneous adipose tissue depth will be measured using the technique described by Martin et al following booking ultrasonography. Measurements will be taken with the participant recumbent and measurements taken approximately 1cm above the umbilicus in triplicate. These measurements will be added to the dataset.

28 weeks: Oral Glucose Tolerance Test: All participants will be invited to attend for a 75g oral glucose tolerance test at 28 weeks gestation as part of their routine clinical care14. Testing will be performed by clinical midwives in the Day Obstetric Unit. The test will take place in the morning following an overnight fast from 10pm the evening before. Maternal weight will be recorded at this visit. Baseline bloods (24mls in total) will be taken for glucose (4mls) and storage (20mls). Following a drink containing 75g glucose, blood will be taken after 60min and 120mins for glucose (4mls) and storage (4mls). Samples for storage will be processed following collection. Glucose will be analysed in the Regional Biochemistry Laboratory immediately.

Plasma glucose results will available within 4 hours of each OGTT. World Health Organisation criteria will be used to diagnose GDM (fasting glucose ≥ 5.1mmol/l; 1-hr ≥ 10.0mmol/l; 2-hr 8.5mmol/l)15. Each woman will be contacted with the results of their OGTT as per our routine practice with immediate referral to the Diabetes Antenatal Clinic for those diagnosed with GDM. Glucose results will be inputted to the study dataset on a daily basis using a unique patient identifier. Samples for storage will be processed as outlined below. Participant weights will also be entered into a database on a daily basis and linked to clinical/biochemical data via a unique patient identifier.

28 weeks: Fetal ultrasound: At the time of their OGTT, participants will also attend the study ultrasonographer for their study ultrasound scan. Abdominal circumference, head circumference, femur length and estimated fetal weight will be measured using the ellipse function on a Voluson E8 ultrasound scanner at the recommended anatomical sites25. The ultrasonographer will be experienced in fetal ultrasound and blinded to early pregnancy HbA1c results. The same scanner will be used for all study participants. Ultrasound measurements will be recorded initially on a study case report form and transferred daily to the electronic study database.

28 weeks: Food Frequency Questionnaire: Each participant will be asked to complete a food frequency questionnaire whilst waiting for blood sampling during their OGTT. This is to evaluate dietary patterns of women with and without GDM and will provide a basis from which future dietary interventions can be formed. The questionnaire used is a validated questionnaire used recently in the Avon Longitudinal Study of Pregnancy and Children (http://www.bristol.ac.uk/alspac)

Delivery: Each participant will continue their usual obstetric care following their 28 week appointment. At the end of the study, obstetric outcome information will be extracted from the Northern Ireland Maternity Information System (NIMATS) and, if necessary, paper records. This will include gestational age at delivery, mode of delivery and the fetal, maternal and early neonatal complications as outlined above in the objectives. Delivery outcomes will be linked to the study data using matched unique participant identifiers.

ELIGIBILITY:
Inclusion Criteria:

-

Age ≥ 18yrs, and at least one of the following NICE risk factors for glucose intolerance:

body mass index ≥ 30kg/m2 a family history of diabetes (first-degree relative) previous macrosomic baby (>4.5kg) minority ethnic family origin with a high prevalence of diabetes

Exclusion Criteria:

- pre-existing type 1 or type 2 diabetes mellitus, a previous history of GDM, booking HbA1c ≥ 48mmol/mol (6.5%), anaemia diagnosed on booking full blood count, booking diagnosis of a multiple pregnancy, use of corticosteroids or metformin within 12 weeks of booking

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women at risk of glucose intolerance/gestational diabetes
Sampling Method: Non-Probability Sample
Enrollment: 1314 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-21 (Actual); Study Completion 2020-08-04 (Actual)

PRIMARY OUTCOMES:
Excessive Fetal Growth | 28 weeks gestation
  Estimated Fetal Weight ≥90th centile
Excessive Fetal Growth | 28 weeks gestation
  Fetal Abdominal Circumference >90th centile

SECONDARY OUTCOMES:
Gestational Diabetes | 28 weeks gestation
  Gestational Diabetes as defined by WHO criteria
Adverse Pregnancy Outcomes | Delivery
  Adverse Outcomes: LGA, SGA, Macrosomia, Preeclampsia, Pregnancy Induced Hypertension, Shoulder Dystocia, Emergency Ceasarean Section

CONTACTS AND LOCATIONS:
Overall Officials: Una Graham, MB BCh BAO, Principal Investigator — Belfast Health & Social Care Trust
Locations (1):
- Royal Jubilee Maternity Service, Belfast, Northern Ireland, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Individual Case Basis